CLINICAL TRIAL: NCT04869371
Title: A Randomized, Controlled, Single Center Clinical Trial to Evaluate the Efficacy and Safety of Neoadjuvant Therapy With Androgen Deprivation Therapy Combined With Docetaxel for High Risk and Very High Risk Prostate Cancer
Brief Title: Androgen Deprivation Therapy Combined With Docetaxel for High Risk Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hongqian Guo (Other)
Responsible Party: Sponsor-Investigator, Hongqian Guo, chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-PC-106
Record Dates: First submitted 2021-04-09; First posted 2021-05-03 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Neoadjuvant Therapy \ High Risk Prostate Cancer \ Docetaxel
MeSH Terms: interventions — Docetaxel; Triptorelin Pamoate; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Androgen Deprivation Therapy with Docetaxel (Experimental): All subjects in this arm will receive luteinizing hormone releasing hormone analogue (LHRHa) plus docetaxel and prednisone, as per standard of care. Triptorelin pamoate (Diphereline) 15mg will be used once per 12 weeks. Docetaxel (75 mg/m2 body surface area) will be administered as intravenous drip every 3 weeks for 6 cycles. Robot assisted radical prostatectomy will be followed in 2 weeks when 24-week treatment cycle is finished.
  Interventions: Drug: Docetaxel injection; Drug: Triptorelin Pamoate for Injectable Suspension; Drug: Prednisone Acetate Tablets
- ADT alone (Active Comparator): All subjects in this arm will receive LHRHa alone for 24 weeks before receiving robot assisted radical prostatectomy. Triptorelin Pamoate 15mg will be administered once per 12 weeks.
  Interventions: Drug: Triptorelin Pamoate for Injectable Suspension

INTERVENTIONS:
Drug: Docetaxel injection — 75 mg/m2 body surface area every 3 weeks for 6 cycles before robot assisted radical prostatectomy
  Arms: Androgen Deprivation Therapy with Docetaxel
Drug: Triptorelin Pamoate for Injectable Suspension — 15mg every 12 weeks
Drug: Prednisone Acetate Tablets — 5 mg oral low dose prednisone, once daily
  Arms: Androgen Deprivation Therapy with Docetaxel

SUMMARY:
This randomized, controlled, single center clinical trial aims to evaluate the efficacy and safety of Androgen Deprivation Therapy Combined with Docetaxel for High Risk Prostate Cancer with a six-month treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 and ≤75 years of age.
* All patients must have a histologically or cytologically diagnosis of prostate cancer and must be eligible for radical prostatectomy.
* All patients must undergo thorough tumor staging and meet one of the following criteria:

  1. multi-parameter MRI or PSMA PET / CT shows clinical staging of primary tumor ≥ T3,
  2. Gleason score of primary tumor ≥ 8, 3.prostate specific antigen (PSA) ≥20 ng/ml.
  3. Eastern Cooperative Oncology Group (ECOG) physical condition score ≤ 1.
  4. Patients must have adequate hematologic function, within 28 days prior to registration as evidenced by: white blood cell (WBC) ≥ 4.0 × 109 /L, platelets≥ 100 × 109 / L, hemoglobin ≥ 9 g / dL, and international normalized ratio (INR) < 1.5.
  5. Patients must have adequate hepatic function, within 28 days prior to registration, as evidenced by: total bilirubin (TBIL)≤1.5 x upper limit of normal (ULN),and SGOT (AST) and SGPT (ALT) ≤ 2.5 x ULN.
  6. Patients must have adequate renal function, within 28 days prior toregistration, as evidenced by serum creatinine ≤2×ULN
* Patients must participate voluntarily and sign an informed consent form(ICF), indicating that they understand the purpose and required procedures of the study, and are willing to participate in. Patients must be willing to obey the prohibitions and restrictions specified in the research protocol.

Exclusion Criteria:

* Patients with prostate having neuroendocrine, small cell, or sarcoma-like features are not eligible.
* Patients with low-risk and medium-risk, localized prostate cancer (the following conditions are met at the same time) are not eligible: multiparameter MRI or PSMA PET / CT shows clinical staging of primary tumor < T3, Gleason score of primary tumor < 8, and prostate specific antigen (PSA) <20 ng/ml.
* Patients with clinical or radiological evidence of extra-regional lymph node metastases or bone metastases or visceral metastases are not eligible.
* Patients who have previously received androgen deprivation therapy (medical or surgical) or focal treatment of prostate cancer or prostate cancer radiotherapy or prostate cancer chemotherapy are not eligible.
* Patients with severe or uncontrolled concurrent infections are not eligible.
* Patients must not have New York Heart Association Class III or IV congestive heart failure at the time of screening. Patients must not have any thromboembolic event, unstable angina pectoris, myocardial infarction within 6 months prior to registration.
* Patients must not have uncontrolled severe hypertension, persistent uncontrolled diabetes, oxygen-dependent lung disease, chronic liver disease, or HIV infection.
* Patients must not have had other malignancies other than prostate cancer in the past 5 years, but cured basal cell or squamous cell skin cancers can be enrolled.
* Patients with mental illness, mental disability or inability to give informed consent are not eligible.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response Rate | up to 8 months
  The proportion of subjects with no morphologically recognizable cancer cell in tumor specimens after radical prostatectomy.
pCR or MRD rate | up to 8 months
  The proportion of patients with pCR or MRD. Pathologic complete response (pCR): defined as no morphologically recognizable cancer cell in tumor specimens after radical prostatectomy.
  Minimal Residual Disease (MRD): defined as residual tumors with maximum diameter of 3 mm or less after radical prostatectomy.

SECONDARY OUTCOMES:
Imaging Response Rate | up to 8 months
  The proportion of subjects whose primary tumor is in complete remission on imaging or residual tumor's maximum diameter is less than 0.5cm.
Rate of Stage Degradation | up to 8 months
  Clinical or pathological stage degradation after neoadjuvant therapy
Rate of Positive Surgical Margins | up to 8 months
  The proportion of subjects with positive surgical margins after radical prostatectomy.
Rate of Complete Serum Remission | up to 8 months
  The proportion of subjects whose PSA is less than or equal to 0.2 ng/ml after 6 months of treatment.
Operative time (min) | 12 month
  The operative time(min) of radical prostatectomy.
Estimated blood loss (ml) | 12 month
  Estimated blood loss (ml) during the process of radical prostatectomy.
Hospital length of stay (day) | 12 month
  The hospitalization time, recorded in day.
Drainage duration (day) | 12 month
  Length of drainage duration, recorded in day.
Incidence of complications (%) | 12 month
  The proportion of subjects who suffer from major complications.
Recovery time of urinary continence (day) | 12 month
  The recovery time of urinary continence (day) after radical prostatectomy, defined as 0 pad/day.
biochemical progression-free survival (bPFS) | 3 years
  Biochemical progression was defined as two consecutive rising PSA values that were above 0.2ng/ml at least one month apart, or starting adjuvant therapy after surgery including radiotherapy, ADT or anti-androgen therapy. The time for bPFS was measured from randomization to biochemical progression or death from any cause.
metastasis-free survival (MFS) | 5 years
  Time from date of randomization to date of evidence of systemic disease on bone scan or cross-sectional imaging.
Serum complete response rate | after 6 month neoadjuvant therapy and before surgery
  Serum complete response rate, defined as the proportion of participants with PSA ≤ 0.1 ng/mL after 6-month neoadjuvant therapy.
Rate of extracapsular extension | 12 month
  The proportion of patients with extracapsular extension on pathologic specimens after neoadjuvant therapy.
Rate of positive lymph node | 12 month
  The proportion of patients with positive lymph node on pathologic specimens after neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, MD, Principal Investigator — Nanjing Drum Tower Hospital, affiliated to medical school of Nanjing University
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhuang J, Wang Y, Zhang S, Fu Y, Huang H, Lyu X, Zhang S, Marra G, Xu L, Qiu X, Guo H. Androgen deprivation therapy plus abiraterone or docetaxel as neoadjuvant therapy for very-high-risk prostate cancer: a pooled analysis of two phase II trials. Front Pharmacol. 2023 Jun 26;14:1217303. doi: 10.3389/fphar.2023.1217303. eCollection 2023. PMID 37435500